CLINICAL TRIAL: NCT03217656
Title: The Jiaxing Birth Cohort in China
Acronym: JBC
Status: Recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Jiaxing Maternity and Child Health Care Hospital (Other); Qingdao University (Other); Westlake University (Other)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Other Study IDs: ZJU_JBC2013013
Record Dates: First submitted 2017-06-18; First posted 2017-07-14 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Childhood Obesity; Anemia; Pregnancy Complications; Pregnancy; Hypertension; Feeding Behavior
MeSH Terms: conditions — Pediatric Obesity; Anemia; Pregnancy Complications; Hypertension, Pregnancy-Induced; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-child birth cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The Jiaxing Birth Cohort (JBC) is the largest prospective cohort study to explore prenatal risk factors, early life feeding practice and growth pattern/ adiposity in Chinese children.Between 1999 and 2013, 338 413 mother-child pairs were recruited in Jiaxing area in south-east China.Children of the recruited women were followed up at 1-2, 3, 6, 9 and 12 months of age, and subsequently followed up every 6 months to 36 months of age (toddler stage), and every year to 6-7 years of age before they went to school (pre-school stage). Follow-up rate was 70.8% at the toddler stage and 68.9% at the pre-school stage up to June 2013.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women came to clinic visit at one of the local hospitals during pregnancy at Jiaxing area
2. Pregnant women were followed up during pregnancy and their children were born alive at local hospital or clinics

Exclusion Criteria:

1. Those who did not want to participant
2. The infant was dead at the birth
3. Those pregnant mothers who dropped out during follow-up at pregnancy or moved out of the Jiaxing area

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Between 1999 and 2013, 363 416 pregnancies were followed from initial registration to the end of the pregnancy, with 25 003 children born to the above women having no further information (registration) after the birth. Therefore, a total of 338 413 live mother-child pairs registered at local clinics, and were enrolled in the Jiaxing Birth Cohort.
  Among the 338 413 children, there were 332 532 singletons, 2883 pairs of twins (n = 5766), 37 pairs of triplets (n= 111), and 1 pair of quadruplets (n = 4).
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 1999-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
overweight and obesity | Up to 6-7 years old for these children
  BMI-z-score was calculated from height and weight. BMI-z-score>1 was defined as overweight/obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Zheng JS, Liu H, Jiang J, Huang T, Wang F, Guan Y, Li D. Cohort Profile: The Jiaxing Birth Cohort in China. Int J Epidemiol. 2017 Oct 1;46(5):1382-1382g. doi: 10.1093/ije/dyw203. No abstract available. PMID 27940484